CLINICAL TRIAL: NCT01340482
Title: A Phase I/II, Open-Label, Repeat-Dose, Dose-Escalation Study of KRN23 in Adult Subjects With X-Linked Hypophosphatemia
Brief Title: A Repeated Study of KRN23 in Adults With X-Linked Hypophosphatemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRN23-INT-001
Record Dates: First submitted 2011-04-15; First posted 2011-04-22 (Estimated); Results first posted 2020-10-26 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: X-linked Hypophosphatemia
Keywords: XLH
MeSH Terms: conditions — Familial Hypophosphatemic Rickets | interventions — burosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KRN23 (Experimental): Escalating doses of KRN23 (0.05, 0.10, 0.30 and 0.60 mg/kg) will be administered SC every 28 days (up to 4 doses)
  Interventions: Drug: KRN23

INTERVENTIONS:
Drug: KRN23 — Subjects will receive escalating doses of KRN23 administered by SC injections every 28-days (up to 4 doses) based on a dosing algorithm and discretion of the investigator and sponsor.

SUMMARY:
The primary purpose of this study is to assess the safety and efficacy of repeated subcutaneous (SC) injections of KRN23 in adult subjects with X-Linked Hypophosphatemia (XLH). A Bone Substudy will evaluate the effects of single-blind KRN23 versus Placebo on bone mineral density and bone quality.

ELIGIBILITY:
Main Inclusion Criteria:

1. 18 years or older
2. Clinical diagnosis of XLH
3. TmP/GFR < 2.0 mg/dL
4. GFR ≥60 mL/min
5. Corrected Ca <10.8 mg/dL
6. A willingness to utilize adequate contraception and not become pregnant[or to have their partner(s) become pregnant] during the study
7. Additional inclusion criteria apply

Main Exclusion Criteria:

1. Have any sign of active infectious disease or have had an infection requiring treatment with antibiotics within 3-weeks of Screening
2. History of known immunodeficiency
3. Pregnant or lactating females subjects or female planning to be become pregnant during the study
4. Receipt of a live (attenuated) vaccine (except for influenza vaccines) within 3-months of Screening, and/or during the study
5. Use of pharmacologic vitamin D metabolite or its analog, phosphate, calcimimetics, and ingestion of aluminum hydroxide antacids within 10-days prior to Screening and/or dosing
6. Use of any supplement containing phosphate, calcium and/or vitamin D within 10-days prior to Screening and/or dosing
7. Condition which could present a concern for either the subject's safety or difficulty with data interpretation
8. Additional exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-04; Primary Completion 2013-05 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Zhang, PhD, Study Director — Kyowa Hakko Kirin Pharma, Inc.
Locations (6):
- United States (5):
  - University of California, San Francisco Medical Center, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Clinical Research Center, Indiana University School of Medicine, Indianapolis, Indiana
  - Duke Clinical Research Unit, Durham, North Carolina
  - University of Texas Health Science Center at Houston, Houston, Texas
- Shriners Hospital for Children - Canada, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Zhang X, Imel EA, Ruppe MD, Weber TJ, Klausner MA, Ito T, Vergeire M, Humphrey J, Glorieux FH, Portale AA, Insogna K, Carpenter TO, Peacock M. Pharmacokinetics and pharmacodynamics of a human monoclonal anti-FGF23 antibody (KRN23) in the first multiple ascending-dose trial treating adults with X-linked hypophosphatemia. J Clin Pharmacol. 2016 Feb;56(2):176-85. doi: 10.1002/jcph.570. Epub 2015 Aug 11. PMID 26073451
- [Derived] Imel EA, Zhang X, Ruppe MD, Weber TJ, Klausner MA, Ito T, Vergeire M, Humphrey JS, Glorieux FH, Portale AA, Insogna K, Peacock M, Carpenter TO. Prolonged Correction of Serum Phosphorus in Adults With X-Linked Hypophosphatemia Using Monthly Doses of KRN23. J Clin Endocrinol Metab. 2015 Jul;100(7):2565-73. doi: 10.1210/jc.2015-1551. Epub 2015 Apr 28. PMID 25919461
- See also: KNR23-INT-002: An Extension Study of KRN23 in Adults With X-Linked Hypophosphatemia — https://clinicaltrials.gov/ct2/show/NCT01571596?term=KRN23-INT-002&draw=2&rank=1

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | KRN23 | Bone Substudy KRN23 | Bone Substudy Placebo
Started | 27 | 1 | 1
Completed | 25 | 1 | 1
Not Completed | 2 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KRN23 | Bone Substudy KRN23 | Bone Substudy Placebo | Total
Number analyzed (Participants) | 27 | 1 | 1 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 26 | 1 | 1 | 28
  >=65 years | 1 | 0 | 0 | 1
Age, Continuous [Median (Full Range); unit: years] | 42 [19 to 66] | 21 [21 to 21] | 28 [28 to 28] | 41 [19 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 1 | 1 | 20
  Male | 9 | 0 | 0 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 26 | 1 | 1 | 28
  Black/African American/African Caribbean | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 1 | 1 | 2
  United States | 27 | 0 | 0 | 27

OUTCOME MEASURES:

1. Primary Outcome: Safety and Efficacy of Repeated SC Injections of KRN23
Description: Safety and efficacy of repeated SC injections of KRN23 from baseline as assessed by serum phosphorus levels,immunogenicity, adverse events and clinically significant changes in vital signs and laboratory testing.
Time Frame: On-Treatment: 6.5 months, 27 total visits
Measure: Count of Participants; unit: Participants
Arm/Group | KRN23 | Bone Substudy KRN23 | Bone Substudy Placebo
Number analyzed (Participants) | 27 | 1 | 1
Participants
  Subjects reporting at least one TEAE | 24 | 1 | 1
  Subjects who died | 0 | 0 | 0
  Subjects reporting SAE other than death | 0 | 0 | 0
  Subjects reporting at least one DLT | 0 | 0 | 0
  Subjects reporting AE leading to discontinuation | 1 | 0 | 0

2. Secondary Outcome: Evaluation of Effect of Repeated SC Injections of KRN23
Description: Effect of repeated SC injections of KRN23, from baseline, on pharmacodynamic parameters including serum phosphorus, sex hormone, bone biomarkers, quality of life assessments and population pharmacokinetics of KRN23 dose levels from cumulative dosing. Summary of serum phosphorus by visit/day is captured below.
Time Frame: On-Treatment: 6.5 months, 27 total visits
Population: Efficacy analysis set: All subjects who received at least 1 dose of KRN23 and completed at least one 28-day post-dose evaluation.
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | KRN23
Number analyzed (Participants) | 26
mg/dL
  Visit 2 (D0)/0 | 1.89 [1.2 to 2.8]
  Visit 3 (D3)/3 | 2.18 [1.5 to 2.9]
  Visit 4 (D7)/7 | 2.20 [1.7 to 3.2]
  Visit 5 (D12)/12 | 2.14 [1.7 to 2.7]
  Visit 6 (D18)/18 | 2.15 [1.7 to 3.0]
  Visit 7 (D26)/26 | 1.96 [1.4 to 2.7]
  Visit 8 (D28)/0 | 1.93 [1.3 to 2.6]
  Visit 9 (D31)/3 | 2.35 [1.5 to 3.3]
  Visit 10 (D35)/7 | 2.45 [1.9 to 3.1]
  Visit 11 (D40)/12 | 2.31 [1.6 to 3.2]
  Visit 12 (D46)/18 | 2.28 [1.3 to 3.0]
  Visit 13 (D54)/26 | 2.15 [1.7 to 3.0]
  Visit 14 (D56)/0 | 2.12 [1.5 to 2.7]
  Visit 15 (D59)/3 | 2.57 [1.7 to 3.8]
  Visit 16 (D63)/7 | 2.85 [1.9 to 3.5]
  Visit 17 (D68)/12 | 2.83 [1.9 to 3.9]
  Visit 18 (D74)/18 | 2.60 [1.6 to 3.5]
  Visit 19 (D82)/26 | 2.33 [1.7 to 3.0]
  Visit 20 (D84)/0 | 2.26 [1.8 to 3.0]
  Visit 21 (D87)/3 | 2.64 [1.9 to 3.6]
  Visit 22 (D91)/7 | 3.03 [2.3 to 3.7]
  Visit 23 (D96)/12 | 2.94 [2.2 to 3.5]
  Visit 24 (D102)/18 | 2.82 [1.7 to 4.0]
  Visit 25 (D110)/26 | 2.54 [1.9 to 3.3]
  End of Study - Visit 26 (D120): number analyzed (Participants) | 25
  End of Study - Visit 26 (D120) | 2.22 [1.6 to 2.9]
  Early Withdrawal: number analyzed (Participants) | 1
  Early Withdrawal | 1.30 [1.3 to 1.3]

3. Other Pre Specified Outcome: Evaluation of Effect of Repeated SC Injections of KRN23 in Bone Substudy
Description: Evaluation of effect of repeated SC injections of KRN23, compared to Placebo on bone mineral density and bone quality.
Time Frame: On-Treatment: 6.5 months, 27 total visits
Population: Subjects randomized to the bone density substudy
Measure: Number; unit: units on a scale
Arm/Group | Bone Substudy KRN23 | Bone Substudy Placebo
Number analyzed (Participants) | 1 | 1
units on a scale | NA — Peripheral quantitative CT and DXA (spine and femur) bone mineral density scans were performed for 2 subjects in the bone substudy. Due to limited sample size for KRN23 and placebo (1 subject each), no meaningful conclusion can be made. | NA — Peripheral quantitative CT and DXA (spine and femur) bone mineral density scans were performed for 2 subjects in the bone substudy. Due to limited sample size for KRN23 and placebo (1 subject each), no meaningful conclusion can be made.

ADVERSE EVENTS:
Time Frame: Subjects were monitored for any untoward medical occurrences from the time of signed ICF through 30 days postdose.
Arm/Group | KRN23 | Bone Substudy KRN23 | Bone Substudy Placebo
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 24/27 | 1/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KRN23 (N=27) | Bone Substudy KRN23 (N=1) | Bone Substudy Placebo (N=1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (4) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (5) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Sensitivity of teeth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0)
Vessel puncture site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 1 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Local swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site urticaria (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (2) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (2) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 7 (8) | 1 (2) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (6) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Ligament pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 1 (7) | 0 (0)
Visual field defect (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 5 (5) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 1 (5)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 1 (4) | 1 (2)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 2 (3) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Only 2 subjects were randomized in and completed the bone substudy. Subsequently, the Sponsor terminated the bone substudy due to slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days